CLINICAL TRIAL: NCT01586130
Title: Assessing the Impact of Isokinetic Muscular Strengthening in Eccentric Mode in the Medical Treatment of Knee Osteoarthritis.
Acronym: ISOGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CHU-0114
Record Dates: First submitted 2012-02-16; First posted 2012-04-26 (Estimated); Last update posted 2024-02-15 (Actual); Status verified 2013-01

CONDITIONS: Unilateral Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Exercise; Isokinetic; Muscle strength; Rehabilitation
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- isokinetic exercises in eccentric mode (Other)
  Interventions: Other: Exercise in eccentric or concentric mode
- isokinetic exercises in concentric mode (Other)
  Interventions: Other: Exercise in eccentric or concentric mode

INTERVENTIONS:
Other: Exercise in eccentric or concentric mode — In this therapeutic field, isokinetic exercises seem to have a better efficiency than other, more frequently used, kinds of exercises such as isometric or isotonic exercises.

SUMMARY:
Knee osteoarthritis (O.A. from now on) is associated to muscular weakness of inferior limbs, especially the quadriceps; leading to disease progression. Advantages of muscular strength training for the treatment of this kind of O.A. is now well established. In this therapeutic field, isokinetic exercises seem to have a better efficiency than other, more frequently used, kinds of exercises such as isometric or isotonic exercises.

Functional impairment caused by knee O.A. is mainly affecting walking. Walking induces muscles to work in eccentric mode.

The hypothesis of this study is that muscular strengthening using isokinetic exercises in eccentric mode would have a more important benefit than isokinetic exercises in concentric mode. Such an hypothesis, if verified, could lead to a better management of rehabilitative knee exercises in the treatment of knee O.A.

DETAILED DESCRIPTION:
Knee osteoarthritis (O.A. from now on) is associated to muscular weakness of inferior limbs, especially the quadriceps; leading to disease progression. Advantages of muscular strength training for the treatment of this kind of O.A. is now well established. In this therapeutic field, isokinetic exercises seem to have a better efficiency than other, more frequently used, kinds of exercises such as isometric or isotonic exercises.

Functional impairment caused by knee O.A. is mainly affecting walking. Walking induces muscles to work in eccentric mode.

The hypothesis of this study is that muscular strengthening using isokinetic exercises in eccentric mode would have a more important benefit than isokinetic exercises in concentric mode. Such an hypothesis, if verified, could lead to a better management of rehabilitative knee exercises in the treatment of knee O.A.

ELIGIBILITY:
Inclusion Criteria:

* Patient male or female, age ranging from 40 to 70 years old
* Patient suffering from one-sided knee O.A. regarding criteria of the American College of Rheumatology (A.C.R.), with radiologic score ranging from 2 to 3 according to the Kellgren & Lawrence classification.
* Patient receiving medical support
* Patient that did not receive any infiltration on knee within two months before randomisation.
* Patient free from any disease that could be a contraindication to the study treatment
* Patient able to understand the protocol and willing to comply with its rules.
* Patient willing to give consent.
* Patient affiliated to the french social secu

Exclusion Criteria:

* Patient carrying prosthesis.
* Patient suffering from inflammatory arthritis, or flare of arthritis.
* Patient suffering from symptomatic patellofemoral osteoarthritis.
* Patient suffering from cardio-vascular or pneumologic disease that could a contraindication to the study treatment.
* Patient suffering from any pathology that could cause muscular weakness (myopathy, neuropathy, hemiplegia...)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-02; Primary Completion 2014-08 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Difference of peak torque of quadriceps | 6 months after treatment start

SECONDARY OUTCOMES:
Walk speed (50 meters and 200 meters) | at day 1, 6 weeks, and 6 months :
Knee pain (via analogic visual scales) | at day 1, 6 weeks, and 6 months
Posture parameters (posturography) | at day 1, 6 weeks, and 6 months
WOMAC Scores | at day 1, 6 weeks, and 6 months
Knee perimeter | at day 1, 6 weeks, and 6 months
Knee range of motion (goniometer) | at day 1, 6 weeks, and 6 months
Kellgren & Lawrence scores | at day 1, 6 weeks, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel COUDEYRE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Jegu AG, Pereira B, Andant N, Coudeyre E. Effect of eccentric isokinetic strengthening in the rehabilitation of patients with knee osteoarthritis: Isogo, a randomized trial. Trials. 2014 Apr 2;15:106. doi: 10.1186/1745-6215-15-106. PMID 24693988